CLINICAL TRIAL: NCT00548678
Title: Open-Label, Randomized, Single-Dose, Four-Treatment Crossover Study to Evaluate Platelet Function in Healthy Adult Males After Administration of IV Diclofenac Sodium, Oral Diclofenac Potasssium, IV Ketorolac Tromethamine, and Acetylsalicylic Acid
Brief Title: Platelet Function and Safety After IV and Oral Diclofenac, IV Ketorolac and Oral Aspirin in Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Javelin Pharmaceuticals (Industry)
Responsible Party: Javelin Pharmaceuticals, Javelin Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DFC-007
Record Dates: First submitted 2007-10-22; First posted 2007-10-24 (Estimated); Last update posted 2008-07-16 (Estimated); Status verified 2008-07

CONDITIONS: Healthy
Keywords: diclofenac, platelet aggregation, ketorolac, aspirin
MeSH Terms: interventions — Ketorolac; Diclofenac; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): intravenous diclofenac sodium
  Interventions: Drug: intravenous diclofenac sodium (DIC075V)
- B (Active Comparator): intravenous ketorolac
  Interventions: Drug: ketorolac
- C (Active Comparator): oral diclofenac (Cataflam)
  Interventions: Drug: oral diclofenac (Cataflam)
- D (Active Comparator): oral aspirin
  Interventions: Drug: aspirin

INTERVENTIONS:
Drug: intravenous diclofenac sodium (DIC075V) — intravenous diclofenac sodium
  Arms: A
Drug: ketorolac — intravenous ketorolac
  Arms: B
Drug: oral diclofenac (Cataflam) — oral diclofenac (Cataflam)
  Arms: C
Drug: aspirin — oral aspirin
  Arms: D

SUMMARY:
This study will assess platelet function and safety in healthy male volunteers following doses of intravenous diclofenac compared to oral diclofenac (Cataflam), intravenous ketorolac and oral aspirin.

DETAILED DESCRIPTION:
The primary objective is to evaluate platelet function following intravenous diclofenac, oral diclofenac (Cataflam), intravenous ketorolac and oral aspirin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects.
* Willing and able to stay at the clinical site for approximately 8 nights over 9 days and to return to the clinic approximately 7 days after discharge.

Exclusion Criteria:

* Bleeding abnormalities or cardiovascular events.
* Known allergy or hypersensitivity to the active compounds or any of the excipients used in the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Area under the platelet closure time curve from 0-6 hours (AUC 0-6 hours) as measured by the PFA-100. | 6 hours

SECONDARY OUTCOMES:
The secondary endpoint is the maximum change from baseline in closure time as measured by the PFA-100. | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Javelin Pharmaceuticals, Study Director — Javelin Pharmaceuticals
Locations (1):
- Comprehensive Phase One, Miramar, Florida, United States